CLINICAL TRIAL: NCT03660072
Title: Empliciti (Elotuzumab) Postmarketing Surveillance in Korean Patients With Multiple Myeloma
Brief Title: Postmarketing Study of Empliciti in Korean Patients With Multiple Myeloma
Status: Withdrawn | Type: Observational
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA204-176
Record Dates: First submitted 2018-08-20; First posted 2018-09-06 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Empliciti combination therapy: Adult patients with a confirmed diagnosis of MM who have received, are currently receiving, or will begin Empliciti combination therapy
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
This study is a regulatory postmarketing surveillance study for Empliciti with a representative sample of the overall Korean multiple myeloma (MM) population.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants who have a confirmed diagnosis of Multiple Myeloma (MM)

Exclusion Criteria:

* Participants who use Empliciti for therapeutic indications which are not approved for Empliciti combination therapy in Korea
* Patients in whom treatment with Empliciti (as clarified in the Korean label) is contraindicated

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean participants with Multiple Myeloma
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01-31 (Estimated); Primary Completion 2022-10-28 (Estimated); Study Completion 2022-10-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of AE's and SAE's | 24 Months

SECONDARY OUTCOMES:
Overall response of Empliciti treatment with lenalidomide and dexamethasone | 24 Months
Incidence of infusion-related reactions associated with Empliciti treatment in combination with lenalidomide and dexamethasone | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Seoul, South Korea

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm